CLINICAL TRIAL: NCT05527106
Title: Evaluation of the Effect of Citicoline (Cebrolux 800 mg) and Docosahexaenoic Acid (DHA) Compound (BrudyPio 1.5 g) on the Visual Function of Patients With Glaucoma With a Pilot Study
Brief Title: Evaluation of the Effect of Citicoline and Docosahexaenoic Acid (DHA) on the Visual Function of Patients With Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Catala de Retina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ICR-14/13
Record Dates: First submitted 2022-08-29; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Glaucoma
Keywords: glaucoma; nutraceuticals; dha (docosahexaenoic acid); citicoline
MeSH Terms: conditions — Glaucoma | interventions — Cytidine Diphosphate Choline; Docosahexaenoic Acids; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Citicoline (Experimental): Cebrolux 800 is a food supplement based on citicoline (163 mg) that also contains vitamin A, E, C and B6.
  Interventions: Dietary Supplement: Citicoline
- Docosahexaenoic Acid (DHA) (Experimental): Brudypio 1.5g is a food supplement based on Omega-3 fatty acid in the form of triglycerides (DHA 70% [350 mg], EPA 8.5%, DPA 6%) that also contains vitamins (A, B1, B2, B3, B6, B9, B12, C, E), carotenoids ( lutein, zeaxanthin, lycopene), glutathione, coenzyme Q10 and minerals (Zn, Se, Cu, Mn).
  Interventions: Dietary Supplement: Docosahexaenoic Acid (DHA)
- Citicoline and Docosahexaenoic Acid (DHA) (Experimental): Cebrolux 800 and Brudypio 1.5g (see above).
  Interventions: Dietary Supplement: Citicoline and Docosahexaenoic Acid (DHA)
- Vitamin C (Experimental): Vitamin C.
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Citicoline — Every subject randomized into this group have to take 2 sachets of Cebrolux 800 (362 mg of citicoline per day), every day, for 3 months.
  Other Names: Cebrolux 800
  Arms: Citicoline
Dietary Supplement: Docosahexaenoic Acid (DHA) — Every subject randomized into this group have to take 3 pills of Brudypio 1.5g (1050 mg of DHA per day), every day, for 3 months.
  Other Names: Brudypio 1.5g
  Arms: Docosahexaenoic Acid (DHA)
Dietary Supplement: Citicoline and Docosahexaenoic Acid (DHA) — Every subject randomized into this group have to take 2 sachets of Cebrolux 800 and 3 pills of Brudypio 1.5g per day, every day, for 3 months.
  Arms: Citicoline and Docosahexaenoic Acid (DHA)
Dietary Supplement: Vitamin C — Every subject randomized into this group have to take 1 pills of Vitamin C (500 mg per day), every day, for 3 months.
  Other Names: L-ascorbic acid
  Arms: Vitamin C

SUMMARY:
Pilot, single-blind, randomized and controlled study to evaluate the changes produced in the visual function of patients with glaucoma after oral administration for 3 months of citicoline and docosahexaenoic Acid (DHA) vs citicoline and docosahexaenoic Acid (DHA) vs vitamin C.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic, primary or secondary, open or closed angle glaucoma, diagnosed by meeting the following criteria:

   * Signs of structural damage: thinning of the optical nerve or peripapillary hemorrhage or decrease in the nerve fiber layer that can be seen by OCT.
   * Signs of functional damage: 3 points outside 95% of the normal limit on the visual field pattern deviation graph.
2. There must be at least 3 reliable visual fields prior to the start of the study.
3. Patients between 50 and 75 years old, homogeneously distributed among the groups.
4. Glaucoma with functional and structural damage.

   * Medium grade, Mean Deviation (MD) between -4 and -20 dB.
   * In at least one eye.

Exclusion Criteria:

1. Treatment with some other vitamin or nutraceutical preparation.
2. Any pathology that can alter the visual field. (Neurological diseases, retinopathies, advanced cataract, patients treated with lyrica (due to the affectation it produces in the visual field)).
3. Hypersensitivity to aspirin. (Cross-allergic reaction has been reported in patients taking citicoline.)
4. Allergic to fish protein.
5. Eye surgery in the 3 months before or during the study.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-03-12 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Effect on Mean Defect (MD) | From Baseline to Month 3.
  Evaluation of changes on the MD (decibels) with study treatment.
Effect on Visual Field Index (VFI) | From Baseline to Month 3.
  Evaluation of changes on the VFI (%) with study treatment.

SECONDARY OUTCOMES:
Evaluation of the changes produced in the intraocular pressure (IOP) | From Baseline to Month 3.
  To compare IOP (mmHg) measurements with study treatment.
Evaluation of tolerance | From Month 1 to Month 3
  Describe the tolerance and the adverse events with study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Anton, MD, PhD, Principal Investigator — Institut Catala de Retina
Locations (1):
- Institut Catala de Retina, Barcelona, Spain